CLINICAL TRIAL: NCT03512093
Title: Born Too Soon in a Resource-limited Setting on the Thailand-Myanmar Border: Can we Improve Care in a Special Care Baby Unit?
Brief Title: Improving SCBU Care for Preterm Babies
Acronym: PretermBabies
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Shoklo Malaria Research Unit (Other)
Responsible Party: Sponsor
Other Study IDs: HCR17005
Record Dates: First submitted 2018-02-19; First posted 2018-04-30 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Preterm Infant; Preterm Birth
Keywords: Preterm Infant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Retrospective chart review
  Interventions: Other: Retrospective chart review
- Focus Group Discussion (FGD) of the medical staff
  Interventions: Other: Focus Group Discussion (FGD) of the medical staff
- Interviews of mothers
  Interventions: Other: Interviews of mothers

INTERVENTIONS:
Other: Retrospective chart review — A retrospective chart review of preterm neonates born in one of the birthing SMRU unit between January 2008 and December 2017 and for whom a medical chart is available. In addition we propose to analyze the growth trajectory, the prevalence of anemia (Hct < 33%) and the level of neurodevelopment achieved in the first year of life reported in the clinical charts of preterm neonates born < 34+0 weeks of gestation.
  Groups: Retrospective chart review
Other: Focus Group Discussion (FGD) of the medical staff — Focus Group Discussion (FGD) of the medical staff working in the SCBU firstly on the benefits and difficulties in using existing guidelines for preterm care and secondly on the feasibility and acceptability of changes in the guidelines 3-6 months after their implementation.
  Groups: Focus Group Discussion (FGD) of the medical staff
Other: Interviews of mothers — Interviews of mothers who delivered preterm neonates (< 37+0 weeks of gestation) to understand the challenges they faced while caring for their child.
  Groups: Interviews of mothers

SUMMARY:
Since 2008, preterm neonates are taking care of in a Special Baby Care Unit (SCBU). Those born less than 34 weeks of gestation are followed-up monthly for one year for monitoring their hematocrit level, growth and development.

Medical chart reviews are useful to evaluate the burden of diseases, characterize care treatment patterns and clinical outcomes by patients' subgroups; ultimately it can help identifying gaps in care pathways thus improving quality of care and ultimately reducing mortality. Medical records of all preterm neonates hospitalized in the SCBU including those followed up during their first year of life are computerized.

The investigators propose to review the clinical charts of the preterm neonates in regards to four main points of care a) feeding, b) infections including early onset of neonatal sepsis, necrotizing enterocolitis and umbilical cord infection, c) body temperature control and d) respiratory distress.

This medical charts review will be complemented by i) focus group discussions (FGD) with the medical staff working in the SCBU on the benefits and difficulties in using the existing guidelines for preterm care and by ii) interviews with mothers who delivered a preterm neonate on their experience in caring for their child and the challenges they faced.

While performing the retrospective part of the project and after discussing the preliminary findings from the medical staff perception of the existing guidelines, the investigators will evaluate the feasibility to implement some additional recommendations to improve preterm birth outcomes based on recent literature and new protocols for resource-limited settings.

DETAILED DESCRIPTION:
This study aims to describe the neonatal clinical outcome of preterm neonates (< 37+0 weeks of gestation) in terms of mortality and prematurity-related morbidity and the growth and neurodevelopment of preterm neonates (< 34+0 weeks of gestation) in the first year of life in order to optimize service delivery for preterm neonates in a resource-constraint setting. The study will consist of 3 parts as follows:

Part A: A retrospective chart review of preterm neonates born in one of the birthing SMRU unit between January 2008 and December 2017 and for whom a medical chart is available. In addition we propose to analyze the growth trajectory, the prevalence of anemia (Hct < 33%) and the level of neurodevelopment achieved in the first year of life reported in the clinical charts of preterm neonates born < 34+0 weeks of gestation.

Part B: Focus Group Discussion (FGD) of the medical staff working in the SCBU firstly on the benefits and difficulties in using existing guidelines for preterm care and secondly on the feasibility and acceptability of the revised guidelines 3-6 months after their implementation.

Part C: Interviews of mothers who delivered preterm neonates (< 37+0 weeks of gestation) to understand the challenges they faced while caring for their child.

This study was funded by Shoklo Malaria Research Unit Core funding (Wellcome Trust). Grant reference number is 220211.

Summary of Results:

Preterm birth is a major public health concern worldwide with the largest burden of morbidity and mortality falling upon the low- and middle-income countries. Evidence-based interventions for preterm neonatal care exist but often meet with barriers to implementation based on constraints in resource-poor settings.

This study summarizes clinical outcomes among preterm neonates born to mothers attending antenatal care at SMRU, regarding four main points of care: feeding, infections, thermal care, and respiratory care. In addition to these clinical outcomes, mixed methods were employed to highlight key implementation outcomes for SCBU care provision in this setting.

Between January 1, 2008, and December 31, 2017, a total of 2319 preterm births were documented, of which, 203 stillbirths were excluded from further analysis. There were 237 deaths documented over the study period, with the proportion of deaths decreasing significantly from 14.4% (144/999) during the early establishment period of SCBU (2008-2011) to 11.0% (66/603) during the expansion of SCBU care to all sites (2012-2014) and to 5.3% (27/514) while the continuum of care was performed more routinely at all sites (2015-2017) (p<0.001). Mortality reduction was observed in all categories of prematurity, with the largest reduction (68%) observed among very preterm neonates (EGA 28-32 weeks). Most deaths (184/237, 77.6%) occurred in the early neonatal period, of which half were within hours of birth (93/184).

Admission for surveillance and further care was routine. Very preterm neonates (EGA 28-32 weeks) remained under observation for nearly three weeks longer than moderate preterm neonates (EGA 33-36 weeks) with a median of 34 days (IQR 20, 49 days) compared to a median of 9 days (IQR 4, 14). Hypothermia (temperature < 36.5ºC) was the most common cause of abnormal body temperature on admission (402/480, 83.8%) independent of prematurity. Nearly one-third of neonates (394/1215, 32.4%) received intravenous antibiotics on admission to SCBU. Duration of oxygen therapy was longer for very preterm (median of 18 days [IQR 10, 32]) compared to moderate preterm neonates (2.5 days [IQR 2-6.5]).

Mothers of neonates (n=9) explained acceptability, satisfaction, and coverage outcomes related to SCBU care. Despite difficult circumstances around access and financial issues, many women realized the need for SCBU care for their newborns. The patient-centered care offset risks associated with both seeking care and the substantial toll that extended hospital stays took on women's personal lives. FGDs with medical staff (n=27) helped explain feasibility, fidelity, and effectiveness outcomes.

Conclusions:

SMRU provides a package of routine and specialized services for antenatal, intrapartum, delivery, postpartum, and newborn care that is facility-based. The package of care for preterm birth and small and sick newborns has evolved over the years and now includes the administration of steroids to women with preterm labor between 27-34 weeks of gestation, maternal antibiotic prophylaxis in case of prolonged rupture of membranes, and diagnosis and treatment of maternal infections The Special Baby Care Units for specialized care of preterm, small, or sick neonates has been equipped with equipment for optimizing respiratory support, phototherapy, feeding, and thermoregulation. The on-site medical staff has been trained in newborn resuscitation and participates in routine exercises based on the Basic Emergency Obstetric & Newborn Care Life Support curriculum. And all these efforts have resulted in a reduction in mortality among all categories of neonates, mostly those very preterms (EGA 28-32 weeks).

However, despite this improvement in survival, interviews and FGDs findings highlighted the barriers in this resource-limited setting and their impact on the feasibility, fidelity, and effectiveness of evidence-based SCBU care. Financial burdens and social issues related to home life were often a pull away from the hospital, hampering the acceptability, appropriateness, and satisfaction mothers felt in accessing clinics or being admitted to the SCBU facility for long periods of time. Medical staff often adapted interventions to fit the financial and environmental constraints imposed by this setting. To further reduce neonatal mortality in preterm neonates there is an urgent need to consider the financial and social constraints on the mothers as well as support to the medical staff that goes beyond improving knowledge.

The final enrolment numbers: Part A: 2116 charts of preterm neonates born to mothers attending ANC at SMRU retrospectively analyzed; 27 participants to FGD and 9 interviews.

ELIGIBILITY:
Inclusion Criteria:

* Part A: Neonatal medical record for preterm neonates (< 37+0 weeks of gestation) in one of the SMRU clinics between January 2008 and December 2017
* Part B: Male or female medical staff (Medics, midwives & nurses) aged 18 years and above, who have been working for SMRU since the introduction of the Special Care Baby Unit (2008-2011) or after its establishment (2012-2017) and have actively cared for preterm newborns. Medical staff (Medics, midwives & nurses) who have provided written informed consent and willing to participate to a Focus Group Discussion
* Part C: Mothers, aged 18 years and above, who have had a preterm newborn (< 37+0 weeks of gestation) admitted in SMRU clinics.

Multigravida or primigravid, presently in the SCBU or already discharged home who willing to discuss the broad topics include caring for the preterm newborn at home. Any mothers will be approached so that responses might provide a comprehensive overview of mothers concerns.

Mothers who have provided written informed consent and willing to participate to an interview

Exclusion Criteria:

• Parts A: Neonatal medical record of neonates < 37+0 weeks of gestation receiving palliative care only.

Neonatal medical record of neonates < 37+0 weeks of gestation born and hospitalized in tertiary hospital.

Neonatal medical record of neonates < 37+0 weeks of gestation born at home and not hospitalized in SMRU clinics during the neonatal period.

Neonatal medical record of neonates < 37+0 weeks of gestation born in SMRU clinics but transferred in tertiary hospital for further neonatal care.

Neonatal medical record of neonates born term (37+0 weeks or more)

* Part B: Medical staff who has never been directly involved in caring for preterm neonates.
* Part C: Mothers aged less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients seeking care to SMRU facilities belong to several distinct ethnic groups present along the Thailand-Myanmar border, mostly from Burman and Karen ethnicity, but also from Mon, Kachin, Shan or Rakhine ethnic background. Medical staff caring for those patients are from the same mixed of ethnic background.
  Part A: All neonates born prematurely (< 37+0 weeks of gestation) in one of the SMRU clinics between January 2008 and December 2017 and for whom a medical record was created between its birth and its first birthday
  Part B: Medical staff directly involved with preterm care
  Part C: Mothers who have delivered a preterm neonate (< 37+0 weeks of estation) in one of the SMRU clinics
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
The neonatal mortality rate of preterm neonates (< 37+ weeks of gestation) expressed in number of newborns dying at less than 28 days of age per 1000 livebirths. | 1 year
The neonatal prematurity-related morbidity rates. | 1 year
  (i.e. necrotizing enterocolitis; sepsis; hypothermia; apnoea of prematurity; respiratory distress syndrome; gastric reflux) expressed as the number of specific-morbidity per number of preterm newborn aged less than 28 days and presented as percentage.
The time lapse between birth and full enteral feeding expressed as mean (SD) days to reach full enteral feeding. | 1 year

SECONDARY OUTCOMES:
The growth trajectory changes during the first year of life of neonates born < 34+0 weeks of gestation expressed as mean (SD) monthly weight/height gain and mean z-scores at end of follow-up. | 1 year
The proportion of anaemia (haematocrit < 33%) during the first year of life of neonates born < 34+0 weeks of gestation. | 1 year
The mean (SD) neurodevelopment score at 6 and 12 month of life of neonates born < 34+0 weeks of gestation. | 1 year
Medical staff and mothers' perception of the difficulties and challenges of caring for preterm neonates analysed by themes and performed using NVivo solfware package. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Shoklo Malaria Research Unit, Mae Sot, Changwat Tak, Thailand

IPD SHARING:
Plan to Share IPD: Yes
All data will be extracted from Microsoft Access databases at SMRU using the existing personal identifier code. Once the link between the paper medical records and the computerized medical records is completed all variables that might identify the patient will be de-identified.
  Participants' data stored in the database for this study may be shared with other researchers to use in the future. However, the other researchers will not be given any information that could identify the participant.
  All audio files will be destroyed when all the transcripts have been completed and verified. De-identified data will be stored digitally as documents that will be password protected. All information will be kept confidential and only research team members will have access to them.
Supporting Information: CSR